CLINICAL TRIAL: NCT00434707
Title: Outcome of Small Pupil Phacotrabeculectomy in Persons With Glaucoma and Cataract
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Aravind Medical Research Foundation (Other)
Other Study IDs: SPTRIPLE0001
Record Dates: First submitted 2007-02-10; First posted 2007-02-13 (Estimated); Last update posted 2007-02-13 (Estimated); Status verified 2007-02

CONDITIONS: Glaucoma; Cataract
Keywords: glaucoma; catarat; small pupils
MeSH Terms: conditions — Glaucoma; Cataract; Miosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Small pupils are not uncommon in situations requiring surgical intervention for glaucoma and cataract. Inadequate binocular view during combined trabeculaectomy and glaucoma surgery needs to be overcome by additional iris manupulations to dilate the pupils which increase the liklihood of inflammation, inraocular pressure rise after surgery and enhnced liklihood of failure of glaucoma surgery. The proposed trial is an observational study to analyse post operative outcome of eyes undrgoing trabeculectomy and phacoemulsification with intraocular lens implantation with small pupils in persons with glaucoma coexisting with cataract.

DETAILED DESCRIPTION:
Small pupils are not uncommon in situations requiring surgical intervention for glaucoma and cataract. Inadequate binocular view during combined trabeculaectomy and glaucoma surgery needs to be overcome by additional iris manupulations to dilate the pupils which increase the liklihood of inflammation, inraocular pressure rise after surgery and enhnced liklihood of failure of glaucoma surgery. The proposed trial is an observational study to analyse post operative outcome of eyes undrgoing trabeculectomy and phacoemulsification with intraocular lens implantation with small pupils in persons with glaucoma coexisting with cataract

ELIGIBILITY:
Inclusion Criteria:

* Individuals with visually significant cataracts and medically uncontrolled primary open angle, angle clsoure, exfolaitive glaucoma

Exclusion Criteria:

* Complicated catracts and secondary glaucoma

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2007-03; Study Completion 2007-12

CONTACTS AND LOCATIONS:
Overall Officials: Ramasami Krishnadas, MD, Principal Investigator — Aravind Eye Hospital